CLINICAL TRIAL: NCT01972321
Title: Integrated Community Case Management of Common Childhood Diseases: Mozambique and Uganda
Brief Title: ICCM of Common Childhood Diseases: Mozambique and Uganda
Acronym: inSCALE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaria Consortium (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University College, London (Other); Karolinska Institutet (Other); Makerere University (Other)
Responsible Party: Principal Investigator, Karin Källander, Senior Research Advisor, Malaria Consortium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OPP1002407; NCT01810055 (obsolete NCT alias)
Record Dates: First submitted 2013-04-22; First posted 2013-10-30 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Malaria; Pneumonia; Diarrhoea
Keywords: Community health worker; Motivation; Performance; Quality of care; Africa
MeSH Terms: conditions — Malaria; Pneumonia; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Technology supported supervision (Experimental): The technology supported supervision intervention will support the CHWs in providing quality case management for the under-fives who suffer from diarrhea, pneumonia and malaria through unlimited communication with their health facility supervisors and colleagues through closed-user-groups. It will enhance timely reporting of patient data and targeted support supervision on the CHWs who need support from their supervisors. With the CHWs receiving the above support and feedback messages, this will potentially increase CHW motivation, performance and retention. Data reported by CHWs can be used by the district planners to forecasting of medicine procurements and react to drug stock-outs or unusual data trends (e.g. disease outbreaks).
  Interventions: Other: Technology supported supervision; Other: Integrated community case management
- Community supported supervision (Experimental): The community supported supervision intervention will set up village health clubs with the aim to improve child health through a community led forum with the CHW as the main focus point. Village health club meetings will provide a forum where CHWs and community members who are part of the club can work together to identify child health and CHW challenges. They will use village networks, knowledge, creativity and other assets.
  Interventions: Behavioral: Community supported supervision; Other: Integrated community case management
- Control arm (Active Comparator): The CHWs in the control arm will be receiving the standard Ministry of Health designed package to integrated community case management support and supervision.
  Interventions: Other: Integrated community case management

INTERVENTIONS:
Other: Technology supported supervision — CHWs will be provided with mobile phones and solar chargers to carry out the following:
  1. Establish closed user groups (CUGs) to enable two-way communication between CHWs and their supervisors free of charge to the users.
  2. Data submission through mobile phones 2.1. receive motivational performance related feedback provided in response. 2.2. Automated messages to supervisors which 2.2.1. Flags problems and strengths/successes identified in CHWs data 2.2.2. Alerting supervisors as to which CHWs require targeted supervision. 2.3. CHWs data summarised in a user friendly format and made accessible to district statisticians
  3. Monthly motivational short message service (SMS) messages provided to CHWs that are locally relevant to CHW work and that are designed to impact positively on CHW performance.
  Arms: Technology supported supervision
Behavioral: Community supported supervision — CHWs will facilitate the clubs using a learning, planning and action cycle. Club members will rank child health challenges faced by their community using picture cards and decide which one to focus on for each cycle. They will discuss solutions, which include supporting CHWs services, and take actions to meet challenges. They will also promote group decision-making and ownership and through this process gain tangible results. Solutions to health challenges developed by club members are a key focus of the village health club approach. Village Health Clubs are based on 5 guiding principles: clubs are open to all, village owned, intended to support CHW work, strength based, and fun and focused.
  Arms: Community supported supervision
Other: Integrated community case management — Implementation of integrated community case management, with provision of training and equipment to CHWs for diagnosis and treatment of malaria, pneumonia and diarrhoea in children less than 5 years of age. Supportive supervision of CHWs will be provided by assigned health facility supervisors.

SUMMARY:
The aim of the inSCALE project is to test the effect of innovative approaches to increase coverage of integrated community case management, which provides community based-care for diarrhoea, pneumonia and malaria, resulting in more children receiving timely and appropriate care for these three most common childhood illnesses

DETAILED DESCRIPTION:
The Innovations at Scale for Community Access and Lasting Effects (inSCALE) project is identifying and documenting limitations to national scale up of Integrated Community Case Management (ICCM) and aims to demonstrate that coverage and impact of government-led ICCM programmes can be extended if innovative solutions can be found for critical limitations. Based on research, three main constraints have been found to limit coverage of community based management of childhood diseases: supervision, motivation and information flow

Potential solutions to the identified constraints have been formulated based on current knowledge and experiences from Malaria Consortium ICCM implementation and other relevant community-based initiatives in both project countries and elsewhere. Extensive formative research was conducted to support the design of innovations aimed to improve motivation and performance of community health workers.

Innovations which have potential to address the project's aims but lack sufficient evidence of impact are being formally evaluated in a randomised control trial. In Mozambique, a technology based intervention is being tested where community health workers (CHWs) are provided with smart phones to programmed with a tool for decision support, immediate feedback and multimedia audio and images to improve adherence to protocols. The tool will also allow CHWs to send key indicators to a server and to keep a register of patients who can be tracked over time. The indicators submitted will be used for performance monitoring of the CHWs by providing automated timely, digestible reports with targeted follow-up actions for CHW supervisors. In Uganda, one technology and one community based intervention are being evaluated over a 12 month period. In the technology intervention, CHWs are given a Java enabled mobile phone through which they can send their weekly reports and drug stocks, receive immediate feedback based on data submission and monthly motivational messages. The phones in both countries also contain innovative tools such as a respiratory timers to support the CHWs in their work. CHWs and their supervisors are on closed user groups in order to increase communication and support. The community intervention is focused on the running of Village Health Clubs. These are designed to be highly participatory with the CHWs in the role of facilitator, aimed at increasing awareness about the CHW role and improving motivation through the support of the community.

Continuous Ministry of Health support for health facilities to provide referral care and equip community health workers with medicines, tools, supervision and training are critical for the success of the project.

ELIGIBILITY:
Inclusion Criteria:

CHWs in districts with ICCM implementation

Exclusion Criteria:

CHWs in districts without ICCM implementation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2289 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Appropriate treatment of malaria, pneumonia and diarrhoea in children under five years of age | 1 year
  Proportion of children under five years of age with symptoms of malaria, pneumonia and diarrhoea who received appropriate treatment

SECONDARY OUTCOMES:
Community health workers with medicine stock-out <1 week each quarter | 1 year
  The proportion of community health workers with medicine stock-out <1 week each quarter

OTHER OUTCOMES:
Community health worker retention | 1 year
  Proportion of community health workers staying in post after 1 year of implementation of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Meek, PhD, Study Director — Malaria Consortium
Locations (2):
- 6 Districts, Inhambane, Mozambique
- 26 Sub-Counties, Hoima, Please Select, Uganda

REFERENCES:
- [Background] Thondoo M, Strachan DL, Nakirunda M, Ndima S, Muiambo A, Kallander K, Hill Z; InSCALE Study Group. Potential Roles of Mhealth for Community Health Workers: Formative Research With End Users in Uganda and Mozambique. JMIR Mhealth Uhealth. 2015 Jul 23;3(3):e76. doi: 10.2196/mhealth.4208. PMID 26206419
- [Background] Kasteng F, Settumba S, Kallander K, Vassall A; inSCALE Study Group. Valuing the work of unpaid community health workers and exploring the incentives to volunteering in rural Africa. Health Policy Plan. 2016 Mar;31(2):205-16. doi: 10.1093/heapol/czv042. Epub 2015 May 22. PMID 26001813
- [Background] Strachan DL, Kallander K, Nakirunda M, Ndima S, Muiambo A, Hill Z; inSCALE study group. Using theory and formative research to design interventions to improve community health worker motivation, retention and performance in Mozambique and Uganda. Hum Resour Health. 2015 Apr 30;13:25. doi: 10.1186/s12960-015-0020-8. PMID 25925007
- [Background] Kallander K, Strachan D, Soremekun S, Hill Z, Lingam R, Tibenderana J, Kasteng F, Vassall A, Meek S, Kirkwood B. Evaluating the effect of innovative motivation and supervision approaches on community health worker performance and retention in Uganda and Mozambique: study protocol for a randomised controlled trial. Trials. 2015 Apr 12;16:157. doi: 10.1186/s13063-015-0657-6. PMID 25873093
- [Background] Hill Z, Dumbaugh M, Benton L, Kallander K, Strachan D, ten Asbroek A, Tibenderana J, Kirkwood B, Meek S. Supervising community health workers in low-income countries--a review of impact and implementation issues. Glob Health Action. 2014 May 8;7:24085. doi: 10.3402/gha.v7.24085. eCollection 2014. PMID 24815075
- [Background] Nanyonjo A, Makumbi F, Etou P, Tomson G, Kallander K; inSCALE Study Group. Perceived quality of care for common childhood illnesses: facility versus community based providers in Uganda. PLoS One. 2013 Nov 7;8(11):e79943. doi: 10.1371/journal.pone.0079943. eCollection 2013. PMID 24244581
- [Background] Kallander K, Tibenderana JK, Akpogheneta OJ, Strachan DL, Hill Z, ten Asbroek AH, Conteh L, Kirkwood BR, Meek SR. Mobile health (mHealth) approaches and lessons for increased performance and retention of community health workers in low- and middle-income countries: a review. J Med Internet Res. 2013 Jan 25;15(1):e17. doi: 10.2196/jmir.2130. PMID 23353680
- [Background] Nanyonjo A, Nakirunda M, Makumbi F, Tomson G, Kallander K, The inSCALE Study Group. Community acceptability and adoption of integrated community case management in Uganda. Am J Trop Med Hyg. 2012 Nov;87(5 Suppl):97-104. doi: 10.4269/ajtmh.2012.11-0763. PMID 23136284
- [Background] Strachan DL, Kallander K, Ten Asbroek AHA, Kirkwood B, Meek SR, Benton L, Conteh L, Tibenderana J, Hill Z. Interventions to improve motivation and retention of community health workers delivering integrated community case management (iCCM): stakeholder perceptions and priorities. Am J Trop Med Hyg. 2012 Nov;87(5 Suppl):111-119. doi: 10.4269/ajtmh.2012.12-0030. PMID 23136286
- [Background] Nanyonjo A, Ssekitooleko J, Counihan H, Makumbi F, Tomson G, Kallander K. Impact of an integrated community case management programme on uptake of appropriate diarrhoea and pneumonia treatments in Uganda: A propensity score matching and equity analysis study. Int J Equity Health. 2015 Sep 4;14:74. doi: 10.1186/s12939-015-0202-y. PMID 26337975
- [Result] Nanyonjo A, Bagorogoza B, Kasteng F, Ayebale G, Makumbi F, Tomson G, Kallander K; inSCALE study group. Estimating the cost of referral and willingness to pay for referral to higher-level health facilities: a case series study from an integrated community case management programme in Uganda. BMC Health Serv Res. 2015 Aug 28;15:347. doi: 10.1186/s12913-015-1019-5. PMID 26315661
- [Derived] Kallander K, Soremekun S, Strachan DL, Hill Z, Kasteng F, Kertho E, Nanyonjo A, Ten Asbroek G, Nakirunda M, Lumumba P, Ayebale G, Bagorogoza B, Vassall A, Meek S, Tibenderana J, Lingam R, Kirkwood B. Improving community health worker treatment for malaria, diarrhoea, and pneumonia in Uganda through inSCALE community and mHealth innovations: A cluster randomised controlled trial. PLOS Digit Health. 2023 Jun 12;2(6):e0000217. doi: 10.1371/journal.pdig.0000217. eCollection 2023 Jun. PMID 37307519
- [Derived] Batura N, Kasteng F, Condoane J, Bagorogosa B, Castel-Branco AC, Kertho E, Kallander K, Soremekun S, Lingam R, Vassall A; inSCALE study group. Costs of treating childhood malaria, diarrhoea and pneumonia in rural Mozambique and Uganda. Malar J. 2022 Aug 20;21(1):239. doi: 10.1186/s12936-022-04254-y. PMID 35987625
- See also: Project website — http://www.malariaconsortium.org/inscale/